CLINICAL TRIAL: NCT03480776
Title: A Randomized Phase II Double-Blind Placebo-Controlled Trial of Acetylsalicylic Acid (ASA) in Prevention of Ovarian Cancer in Women With BRCA 1/2 Mutations (STICs and STONEs)
Brief Title: ASA in Prevention of Ovarian Cancer (STICs and STONEs)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Apotex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OV25
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer Prevention
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylsalicylic Acid (ASA) (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Sham Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid — 81 mg PO daily or 325 mg PO daily
  Other Names: ASA
  Arms: Acetylsalicylic Acid (ASA)
Other: Placebo — One tablet PO daily
  Arms: Placebo

SUMMARY:
While ASA is not a cancer medication, research suggests that taking ASA reduces the probability of getting many types of cancer because of its anti-inflammatory action. Inflammation in the ovaries during ovulation is thought to contribute to the development of ovarian cancer, and, because ASA is an anti-inflammatory medication, it may help to prevent it.

DETAILED DESCRIPTION:
The standard or usual treatment for women with a high risk gene mutation, BRCA1 or BRCA2, is to have risk-reducing surgery to remove the fallopian tubes and ovaries (bilateral salpingo-oophorectomy or bilateral salpingectomy inclusive of fimbria) after they have decided not to have more children naturally.

Acetylsalicylic Acid (ASA) is a safe, well tolerated drug taken by mouth. ASA has been available for over 100 years and has been used mainly to relieve fever and pain, but also as an anti-inflammatory medication in order to reduce inflammation (swelling).

ELIGIBILITY:
Inclusion Criteria:

* Previously documented germline BRCA1/2 pathogenic mutation or likely pathogenic variant based on the ACMG 2015 guidelines
* Risk-reducing surgery (bilateral salpingo-oophorectomy or bilateral salpingectomy inclusive of fimbria) scheduled for within 6 months to 2 years after the date of randomization as standard of care, for women who have completed their families
* ECOG performance status 0 or 1
* Age ≥ 18 years old
* Subject is able (i.e. sufficiently literate) and willing to complete the Credibility/Expectancy questionnaire in English or French.
* Subject consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each subject must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Subjects must be accessible for treatment and follow up. Subjects randomized on this trial must be treated and followed at the participating centre.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days after subject randomization
* Women of childbearing potential must have agreed to use a highly effective contraceptive method for the duration of the study treatment and for 30 days post last dose of study medication

Exclusion Criteria:

* Subjects with history of other malignancies, except:

  * adequately treated non-melanoma skin cancer;
  * curatively treated in-situ cancer of the cervix;
  * previously diagnosed (at any point) breast cancer, treated with curative intent; prior chemotherapy is allowed and the last dose must be ≥ 12 months prior to randomization; endocrine therapy for breast cancer is allowed at any time.
  * other solid tumours curatively treated with no evidence of disease for > 5 years.
* Subjects who have been treated with any PARP-inhibitors (e.g. olaparib) at any time.
* Subjects with active bleeding or bleeding diathesis.
* Subjects with active peptic ulcer.
* Subjects with renal, hepatic or congestive heart failure.
* Subjects with concurrent use of anti-coagulants and/or anti-platelet agents.
* Subjects with prior bilateral salpingectomy.
* Subjects with history of chronic daily use of ASA or NSAIDs.
* Subjects with intolerance of ASA including subjects with a history of asthma induced by salicylates or substances with a similar action, notably non-steroidal-anti-inflammatory drugs.
* Ongoing or planned pregnancy.
* Subjects who are breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 117 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of pre- & malignant lesions found during prophylactic risk reduction surgery using a stratified Cochran-Mantel-Haenszel test | 5 years

SECONDARY OUTCOMES:
Acceptance of the ASA intervention from the self-report Credibility/Expectancy Questionnaire | 5 years
Compliance of taking ASA by serum monitoring | 5 years

OTHER OUTCOMES:
Compliance of taking ASA by evaluation of treatment completion rates | 5 years
Compliance of taking ASA by reasons for early discontinuation of protocol intervention. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Study Chair — Univ. Health Network-OCI/Princess Margaret Hospital, Toronto, ON Canada; Stephanie Lheureux, Study Chair — Univ. Health Network-OCI/Princess Margaret Hospital, Toronto, ON Canada
Locations (17):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Peter McCallum Cancer Institute, Melbourne, Victoria
  - King Edward Memorial Hospital, Subiaco, Western Australia
  - St John of God Subiaco, Subiaco, Western Australia
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Clinical Research Unit at Vancouver Coastal, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre, Kingston, Ontario
  - North York General Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No